CLINICAL TRIAL: NCT03957317
Title: Improving Sleep Quality and Satisfaction for Postoperative Plastic Surgery Flap Patients in the CUH SICU
Brief Title: Improving Sleep Quality in Flap Patients in the SICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Bryan Romito, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU082017-007
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Sleep Deprivation
Keywords: Surgery; Postoperative sleep deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Ear Protective Devices

STUDY DESIGN:
Intervention Model Description: Randomized, controlled study comparing effects of wearing eye masks and ear plugs for sensory deprivation against the standard-of-care (no treatment). Primary outcome is measuring difference between RCSQ scores (sleep quality survey).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects in this group do not receive an eye mask or ear plugs, and receive standard of care (including pain control modalities). The subjects will receive a Richards-Campbell Sleep Questionnaire (RCSQ) survey for each night they spend in the Surgical ICU, as well as a modified Family Satisfaction in the Intensive Care Unit (FS-ICU) survey upon discharge from the ICU.
- Intervention (Experimental): Subjects in this group receive an eye mask and ear plugs in addition to standard of care for pain control. The subjects will receive a Richards-Campbell Sleep Questionnaire (RCSQ) survey for each night they spend in the Surgical ICU, as well as a modified Family Satisfaction in the Intensive Care Unit (FS-ICU) survey upon discharge from the ICU.
  Interventions: Other: Eye mask and ear plugs

INTERVENTIONS:
Other: Eye mask and ear plugs — Subjects receive one pair of eye mask and ear plugs during their stay in the surgical ICU.
  Arms: Intervention

SUMMARY:
This investigation will be a randomized interventional prospective quality improvement study. Patients undergoing plastic surgery with flap procedures (n =123) will be randomized to evaluate the effect of the implementation bundle for sleep quality improvement in the surgical intensive care unit (SICU). Roughly one half of the patients (n =62) will be randomized to the intervention group. This group will receive the intervention bundle which consists of providing ear plugs and eye masks to patients and their family members. Roughly one half of the patients (n =62) will be randomized to the control group. This group will receive "usual care", which does not include ear plugs or eye masks and lacks specified times for laboratory draws and imaging studies. For each of the two groups, the investigators will collect Richards-Campbell Sleep Questionnaire (RCSQ) scores, Confusion Assessment Method for the ICU (CAM-ICU) scores, and modified Family Satisfaction in the Intensive Care Unit (FS-ICU) scores. The investigators will administer the RCSQ to these patients following every night they spend in the SICU and the FS-ICU questionnaire immediately prior to their discharge from the ICU.

DETAILED DESCRIPTION:
Patients will be identified during their presurgical clinic visit or anesthesia preoperative clinic visit for eligibility. The electronic medical record (Epic) will also be used for prescreening of potential study participants by reviewing the clinic visit daily schedule or operating room schedule. Then patient charts will be reviewed for initial data collection to determine the eligibility of potential subjects with the use of a HIPAA waiver form.

A discussion of risks, benefits, and alternatives will be performed. Following the discussion, informed written consent for clinical care and participation in the study will be obtained.

Roughly one half of the patients (n =62) will be randomized to the intervention group. This group will receive the intervention bundle which consists of providing ear plugs and eye masks to patients and their family members. Roughly one half of the patients (n =62) will be randomized to the control group. This group will receive "usual care", which does not include ear plugs or eye masks and lacks specified times for laboratory draws and imaging studies. For each of the two groups, the investigators will collect RCSQ scores, CAM-ICU scores, and modified FS-ICU scores. The investigators will administer the RCSQ to these patients following every night they spend in the SICU and the modified FS-ICU questionnaire immediately prior to their discharge from the ICU. The RCSQ is a short, 5-question, validated survey instrument for measuring sleep quality in ICU patients. The FS-ICU is a short, validated survey instrument for measuring family satisfaction with care and decision making in the ICU. The modified version is more focused on satisfaction of the patient rather than their family member(s). The CAM-ICU is a validated screening test for delirium, and scores are currently charted in the electronic medical record (EMR) as a part of routine monitoring in the SICU. The anticipated length of time for the project is 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age ≥ 18 years
* Individuals undergoing plastic surgery flap procedures requiring hourly monitoring

Exclusion Criteria:

* Pregnancy
* Incarceration
* Diagnosis of obstructive sleep apnea
* Diagnosis of insomnia or other sleep disturbance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Improvement in Richards-Campbell Sleep Questionnaire (RCSQ) scores | 2 days from ICU admission
  The Richards-Campbell Sleep Questionnaire (RCSQ) is a 5-item questionnaire used to evaluate perceived sleep depth, sleep latency, number of awakenings, efficiency, and sleep quality. Each RCSQ question is measured on a 0 (minimum) to 100 (maximum) visual-analogue scale, with higher scores representing better sleep. The primary outcome measure is a 25% increase in median RCSQ scores from the control group.

SECONDARY OUTCOMES:
Improvement in overall modified Family Satisfaction in the Intensive Care Unit (FS-ICU) survey scores | 2 days from ICU admission
  The Family Satisfaction in the Intensive Care Unit (FS-ICU) questionnaire is a reliable and valid 34-item tool used to measure family satisfaction with care and decision-making in the ICU. Each question is completed using a 5-point Likert scale where 1 = excellent, 2 = very good, 3 = good, 4 = fair, 5 = poor, and 6 = not applicable. A modified version of the FS-ICU survey used in the present study includes 14 questions and contains only questions directed toward the patient and not family members. Overall satisfaction score is calculated as the mean of the 14 items, with lower scores indicating greater satisfaction. A secondary outcome measure is to determine the difference in overall modified FS-ICU scores between control and intervention groups.
Improvement in positive Confusion Assessment Method for the ICU (CAM-ICU) scores | 2 days from ICU admission
  The Confusion Assessment Method for the ICU (CAM-ICU) is a valid and reliable delirium monitoring instrument for ICU patients. It tests for the presence of alteration in mental status, inattention, altered level of consciousness, and disorganized thinking. The presence of both altered mental status and inattention along with either altered consciousness or disorganized thinking corresponds to a positive CAM-ICU result, and delirium is present. If these criteria are not met, then CAM-ICU is considered negative, and delirium is absent. A secondary outcome measure is to determine the difference in positive CAM-ICU results between control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan T Romito, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified aggregate data can be shared with other researchers at this time.

REFERENCES:
- [Derived] Obanor OO, McBroom MM, Elia JM, Ahmed F, Sasaki JD, Murphy KM, Chalk S, Menard GA, Pratt NV, Venkatachalam AM, Romito BT. The Impact of Earplugs and Eye Masks on Sleep Quality in Surgical ICU Patients at Risk for Frequent Awakenings. Crit Care Med. 2021 Sep 1;49(9):e822-e832. doi: 10.1097/CCM.0000000000005031. PMID 33870919